CLINICAL TRIAL: NCT02986620
Title: Italian Registry on the Prevalence of IDH1/IDH2 Mutations in Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: AML1516
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2022-01-04 (Actual); Status verified 2021-09

CONDITIONS: AML, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AML patients: Adult AML patients with the IDH mutation test performed at diagnosis or relapse until January 31st, 2019.
  Interventions: Genetic: IDH mutation test performed at diagnosis or relapse until January 31st, 2019.

INTERVENTIONS:
Genetic: IDH mutation test performed at diagnosis or relapse until January 31st, 2019. — Observation of the test result.

SUMMARY:
This is a study where there are no interventions planned. Investigators will only collect data already in the patient's history and analyze it. Particularly, we are interested in molecular data from AML patients.

This means that patients will follow their regular diagnostic and clinical practice. The analyses will be conducted according to the routine diagnostic and clinical practice as well and no additional blood withdrawal will be performed.

DETAILED DESCRIPTION:
The study will be conducted as follows:

1. Retrospective phase clinical and molecular data of patients analyzed for IDH1/2 mutations will be retrospectively collected in the centers that have already introduced IDH1/2 mutational screening in their practice from cases collected according to standard procedure (Ficoll and lysis in RLT buffer).
2. Prospective phase: each participating center already performing IDH1/2 mutational status on samples of their AML patients at diagnosis or relapse - on freshly isolate mononuclear cells from bone marrow and/or peripheral blood using Ficoll density gradient preparation - will prospectively collect the clinical and molecular data.

ELIGIBILITY:
Inclusion criteria:

* Signed written informed consent according to ICH/EU/GCP and national local laws (if applicable);
* AML patients;
* Age ≥18;
* IDH mutation test performed at diagnosis or relapse until January 31st, 2019.

Exclusion criteria:

* AML M3 subtype according to the FAB classification;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult AML patients
Sampling Method: Non-Probability Sample
Enrollment: 388 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
Number of patients with the IDH mutations in AML at initial diagnosis. | At two years from study entry.
Number of patients with the IDH mutations in AML at relapse. | At three years from study entry.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Martinelli, Study Chair — Department of Experimental, Diagnostic and Specialty Medicine, University of Bologna; Maria Teresa Voso, Study Director — U.O.C. Ematologia Dipartimento di Medicina, Policlinico Tor Vergata of Rome
Locations (24):
- Italy (24):
  - Aon Ss. Antonio E Biagio E C. Arrigo - Alessandria - Soc Ematologia, Alessandria
  - Aou Consorziale Policlinico - Bari - Uo Ematologia Con Trapianto, Bari
  - Aou Di Bologna - Policlinico S. Orsola-Malpighi - Uoc Ematologia, Bologna
  - Istituto di Ematologia "Lorenzo e A. Seragnoli" - Università degli Studi di Bologna - Policlinico S. Orsola - Malpighi, Bologna
  - Asl Brindisi, Ospedale 'Perrino' - Brindisi - Uo Ematologia, Brindisi
  - I.R.S.T. Srl Irccs - Meldola - Sc Oncologia Medica, Meldola
  - AOU Policlinico G. Martino, Messina
  - Asst Grande Ospedale Metropolitano Niguarda - Milano - Sc Ematologia, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico UOC Oncoematologia- Padiglione Marcora 2° piano, Milan
  - Irccs Ospedale S. Raffaele - Milano - Uo Oncoematologia, Milan
  - Istituto Europeo Di Oncologia Irccs - Milano - Divisione Di Oncoematologia, Milan
  - UO Ematologia _AOU Policlinico di Modena, Modena
  - Università degli Studi di Padova - Ematologia ed Immunologia Clinica, Padua
  - Ao Ospedali Riuniti Villa Sofia Cervello - Palermo - Uo Ematologia Con Utmo, Palermo
  - AU Policlinico "Paiolo Giaccone", Palermo
  - Aou Di Parma - Sc Ematologia E Centro Trapianti Midollo Osseo, Parma
  - Sezione di ematologia ed immunologia - Clinica Ospedale S. Maria della Misericordia, Perugia
  - Asl Di Piacenza, Ospedale "Guglielmo Da Saliceto" - Ematologia E Centro Trapianti, Piacenza
  - IFO Istituto Nazionale Tumori Regina Elena, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A.Gemelli, Roma
  - Università degli Studi - Policlinico di Tor Vergata, Roma
  - Università degli Studi - Policlinico Tor Vergata, Rome
  - Ente Ecclesiastico Casa Sollievo Della Sofferenza - San Giovanni Rotondo - Ematologia, San Giovanni Rotondo
  - Asui Di Udine - Presidio Ospedaliero "Santa Maria Della Misericordia" - Clinica Ematologica, Udine

IPD SHARING:
Plan to Share IPD: No